CLINICAL TRIAL: NCT07068633
Title: Korea VHD Echo Study: Surveillance of Aortic, Mitral & Tricuspid Patients - Insights From Real-world Practice
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-1451
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Mitral Valve Prolapse; Tricuspid Valve Insufficiency; Rheumatic Heart Disease; Aortic Diseases
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Mitral Valve Prolapse; Tricuspid Valve Insufficiency; Rheumatic Heart Disease; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aortic petients: Primary focus is aortic stenosis patients; secondary focus is aortic regurgitation.
- Mitral Patients: Primary focus is Degenerative Mitral Regurgitation patients; secondary focus is Functional Mitral Regurgitation.
- Tricuspid Patients: Primary focus is Tircuspid Regurgitation patients

SUMMARY:
Valvular heart disease (VHD) is a growing public health concern globally, with increasing disease burden and rising interest in advanced treatment strategies such as transcatheter interventions. However, there remains a significant lack of real-world data regarding echocardiography practices, disease prevalence and progression, referral patterns, and treatment pathways. Addressing these gaps is critical for improving patient care and informing clinical decision-making.

South Korea provides a unique opportunity to conduct a nationwide retrospective echocardiographic study due to its advanced healthcare infrastructure, high patient volume, and strong tradition in clinical research. The current study aims to evaluate the real-world burden and clinical journey of patients with moderate or severe valvular disease over a 10-year period, based on echocardiographic and electronic medical record (EMR) data collected from multiple tertiary centers across the country.

DETAILED DESCRIPTION:
This is a multicenter, retrospective observational study conducted using data from January 1, 2010 to December 31, 2020. The study will include adult patients (≥18 years old) who underwent at least two transthoracic echocardiograms during the study period. Eligible patients will be identified consecutively from each participating institution's echocardiographic and EMR databases. Patients with moderate or severe valvular heart disease (VHD), as defined by guideline-based echocardiographic criteria, will be included in the final analysis.

Patients with congenital heart disease, previous valve surgery at baseline, or incomplete clinical or imaging data will be excluded. The data collected will include demographics, comorbidities, echocardiographic parameters, and clinical outcomes such as mortality and treatment interventions. Particular attention will be paid to disease severity at baseline, rate of progression (from mild to severe), and time to treatment. Treatment patterns, including referral to surgery or transcatheter valve interventions (e.g., TAVI), will also be explored.

Sampling will follow a non-probability, consecutive patient sampling approach, as patients are retrospectively identified based on predefined eligibility criteria. The final sample size is estimated based on precedent data from a previous Korean VHD study that included ~4,000 patients over a 2-month period across 45 centers. Given the 10-year study duration and the number of participating institutions, a larger and more comprehensive sample is expected in this study.

ELIGIBILITY:
Inclusion Criteria:

* Period: 2010.1.1~2020.12.31
* Age > 18 years
* Moderate or severe native VHD (AS, AR, MR and TR)
* Perform echocardiography more than twice

Exclusion Criteria:

* Poor image of echocardiography
* Follow up loss

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study includes adult patients (≥18 years) diagnosed with moderate or severe valvular heart disease (VHD) between January 1, 2010, and December 31, 2020, at tertiary hospitals in South Korea. Eligible patients must have undergone at least two transthoracic echocardiograms. Patients will be identified consecutively from echocardiographic and electronic medical record (EMR) databases. Exclusion criteria include congenital heart disease, prior valve surgery at baseline, and incomplete imaging or clinical data. Patients will be classified by valve type (aortic stenosis, aortic regurgitation, mitral regurgitation, tricuspid regurgitation), severity (moderate vs. severe), and etiology (degenerative, rheumatic, endocarditis, etc.). Demographic information such as age, sex, and comorbidities will be collected. The estimated sample size is expected to exceed 10,000 patients based on the number of participating centers and the 10-year study period.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Moderate and Severe Valvular Heart Disease (VHD) | January 1, 2010 - December 31, 2020
  Evaluate the prevalence of moderate and severe VHD (including AS, AR, MR, and TR) based on echocardiographic findings and diagnostic records during the study period.
Etiological Classification of Aortic Stenosis (AS) | January 1, 2010 - December 31, 2020
  Classify AS cases retrospectively into degenerative, bicuspid, rheumatic, infective endocarditis, or aortopathy based on clinical records and imaging data.
Etiological Classification of Aortic Regurgitation (AR) | January 1, 2010 - December 31, 2020
  Categorize AR patients according to underlying causes: degenerative, bicuspid, rheumatic, infective endocarditis, or aortopathy.
Etiological Classification of Mitral Regurgitation (MR) | January 1, 2010 - December 31, 2020
  Retrospectively classify MR into primary MR (degenerative, mitral valve prolapse, rheumatic, endocarditis) and secondary MR (ventricular functional MR, atrial functional MR).
Classification of Tricuspid Regurgitation (TR) | January 1, 2010 - December 31, 2020
  Classify TR cases into primary and secondary based on echocardiographic findings and clinical context.
Disease Progression and Treatment Pathway | January 1, 2010 - December 31, 2020
  Analyze the time course of VHD progression from mild to moderate to severe and track the time to intervention (surgical or transcatheter) using retrospective patient records.

SECONDARY OUTCOMES:
All-Cause and Cardiovascular Mortality | From initial diagnosis to date of death or last follow-up (within 2010-2020)
  Assess the incidence of all-cause mortality and cardiovascular-specific mortality among patients with valvular heart disease, using hospital records and national death registry data (if available).
Treatment Pathway by Disease Severity | From initial diagnosis to date of death or last follow-up (within 2010-2020)
  Evaluate how the treatment approach (medical management, surgical valve repair/replacement, or transcatheter intervention) varies according to disease severity (mild, moderate, severe) across different types of VHD.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided